CLINICAL TRIAL: NCT05936437
Title: An Open-label Study Evaluating the Clinical Benefits and Safety of Combined Polynucleotides and Hyaluronic Acid - Newest - for Acne Scars Treatment
Brief Title: Clinical Benefits and Safety of Combined Polynucleotides and Hyaluronic Acid - Newest - for Acne Scars Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEW-ACT-22
Record Dates: First submitted 2023-06-13; First posted 2023-07-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Atrophic Scar
Keywords: Post-acne atrophic scars; Polynucleotides; Hyaluronic acid; Mastelli; Acne scars; Newest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Eligible subjects aged 20 to 60 years and in good general health, with grade 3 to 4 moderate-to-severe atrophic post-acne scars according to the Goodman Baron classification
  Interventions: Device: Subjects treated with Newest medical device

INTERVENTIONS:
Device: Subjects treated with Newest medical device — Newest is a sterile, non-pyrogenic, viscoelastic gel for single use for intradermal infiltrations. Newest is a medical device containing 2ml of the original association of polynucleotides (10mg/ml) and hyaluronic acid (10mg/ml).
  Total number of treatments will consist in 4 Newest administrations: at T0 - basal, at T1- 2 weeks, at T2 - 4 weeks, at T3- 6 weeks.

SUMMARY:
This clinical study wants to evaluate the efficacy and safety of a medical device combining "Polynucleotide Highly Purified Technology" (PN-HPT™) and hyaluronic acid (Newest-Mastelli S.r.l) for treating moderate-to-severe atrophic post-acne scars.

DETAILED DESCRIPTION:
This is a prospective, open label study aimed to evaluate efficacy and safety of Newest in facial acne scars treatment. The study will be conducted at Fatebenefratelli Hospital in Rome (Italy). All procedures have to be conducted in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration of 1975, as revised in 2000 and 2008.

A subject will be involved in the study for 6 months and photographs and instrumental assessment (Antera 3 D) will be performed at 1 months, 2 months, 3 months and 6 months after first treatment administration; results will be compared with basal line evaluation (T0).

The sample size of 30 patients has been selected, based on the previous clinical results obtained from a "Preliminary Prospective and Randomized Study of Highly Purified Polynucleotide vs Placebo in Treatment of Moderate to Severe Acne Scars". This sample size combined with this study model is statistically sufficient to provide robust estimation of the primary endpoint.

The study primary objective is to show the clinical improvement in acne facial scars treated with Newest.

The primary end-point of the study is the variation of post-acne scars characteristics evaluated through the Goodman Baron scale at follow up visits F.U. 3 and F.U. 6 versus baseline visit (T1). At the end of follow-up, an average reduction of at least two points of the Goodman score versus baseline will be considered as a positive outcome.

A descriptive statistical analysis will illustrate the percentage of patients with different score variation versus basal line.

The secondary objectives of the study are the improvement of the skin quality and the safety of the investigational device; the secondary end-points are:

* Centralized evaluation of the photos of scars, taken pre- and post-treatment and evaluated by a blinded investigator. Optionally the differences pre- and post-treatment in skin roughness, texture (elasticity/hydration), colors/evenness, vascular features, and pore dimensions could be also evaluated by means of 3D pictures (Antera 3D® or QuantifiCARE®).
* Aesthetic improvement of depressed facial atrophic scars using the "Global Aesthetic Improvement Scale" (GAIS) performed by both the patient and the investigator15; the percentage of questionnaire score improvement ≥ 2 between the two follow up visits will be considered of a clinical significance.
* Adverse events (AE) will be monitored throughout the trial. A safety assessment has to be conducted by the investigator at each scheduled visit. The intensity (mild/moderate/severe) will be assessed according to the investigator's judgement. If a patient drops out of the study, the possible reasons for drop-out, including no improvement in the scar, or occurrence of unacceptable signs/symptoms, need to be documented.

All the screened patients at the baseline visit (T0), after checking the inclusion/exclusion criteria, will be prospectively randomized in the clinical study. The Investigator has to grade the post-acne scar's severity according to the "Goodman Baron classification". The eligible patient will undergo the first injection with the study medical device and the investigator shall evaluate the clinical result by the Goodman score. At follow up visits the patient and the investigator have to judge the aesthetic improvement of scars by checking the GAIS questionnaire.

A total of 4 administrations of the investigational product are scheduled: at the baseline visit (T1), at T2, T3 and T4, with an interval of 2 weeks from each other. The clinical evaluation (Goodman score) has to be performed in addition to the basal visit (T1) also after 3 and 6 months of follow-up respectively.

Standardized photographs shall be taken prior to the first injection of the study product and at every study visit in order to document treatment effect. A reference basal photo should be taken of each patient, with a snapshot of the facial region most damaged by the acne scars. A service basal photo on which the shooted damaged facial area is marked out should be the reference photo for further evaluations.

Note that no covering make-up should be used on the photographs. Each Investigator and other study site personnel designated to take photographs shall be thoroughly trained in the photographic equipment and techniques before study start, if applicable.

Photographs shall be taken at the baseline visit before treatment (T1). If the photographs are considered good quality, the Investigator may proceed with treatment of the subject; if the photographs are considered not good enough, the photography shall be repeated.

All snapshot must be taken against a neutral background and artificial light only, in same circumstances (same perspective/angle, same distance) and ideally with the same camera (usually using a 5 mega pixel camera and analyzed as for color and pigmentation by a computer program).

The subject should keep the eyes closed during photography and shall have a neutral facial expression.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, with age ≥ 20 and ≤ 60 years with an approximately symmetric number of atrophic acne scars on the whole face;
2. Subject presenting a grade 3 to 4 according to Goodman classification corresponding to moderate-to-severe atrophic post-acne facial scars;
3. Scar lesions have not be active
4. Subject who never underwent surgical or laser face treatment for acne scars;
5. Subjects with prior administration of oral steroids and/or isotretinoin should have interrupted this therapy at least 6 months before study kick off.
6. Subject who agree to discontinue all dermatological treatment and procedures during the study;
7. Subject willing to provide signed informed consent to clinical investigation participation;
8. Subject able to communicate adequately with the Investigator and to comply with the requirements for the entire study

Exclusion Criteria:

1. Patients younger than 20 or older than 60 years;
2. Subjects with mild atrophic acne scars according to the Goodman classification (grade 1-2);
3. Pregnancy or breastfeeding women;
4. Systemic or local illnesses that might affect wound healing
5. Severe solar elastosis or scarring;
6. Concomitant intake of anticoagulant or antiplatelet medications;
7. Subjects who have followed a washout period of 2 weeks from topical corticosteroids, antibiotics, benzoyl-peroxide, azelaic acid, hydroxy acids, topical retinoids;
8. History of autoimmune disease or chronic drug or alcohol abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Goodman Baron score | 6 months
  The primary end-point of the study is the blinded assessment of variations of scar characteristics evaluated through the Goodman Baron score at scheduled visits versus baseline visit (T1)

SECONDARY OUTCOMES:
Skin quality difference | 6 months
  Centralized evaluation of the photos of scars, taken pre- and post-treatment and evaluated by a blinded investigator. Optionally the differences pre- and post-treatment in skin roughness, texture (elasticity/hydration), colors/evenness, vascular features, and pore dimensions could be also evaluated by means of 3D pictures (Antera 3D® or QuantifiCARE®).
Global Aesthetic Improvement Scale | 6 months
  Aesthetic improvement of depressed facial atrophic scars using the "Global Aesthetic Improvement Scale" (GAIS) performed by both the patient and the investigator; the percentage of questionnaire score improvement ≥ 2 between the two follow up visits will be considered of a clinical significance
Adverse events (AE) | 6 months
  Adverse events (AE) will be monitored throughout the trial. A safety assessment has to be conducted by the investigator at each scheduled visit. The intensity (mild/moderate/severe) will be assessed according to the investigator's judgement. If a patient drops out of the study, the possible reasons for drop-out, including no improvement in the scar, or occurrence of unacceptable signs/symptoms, need to be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bartoletti, MD, Principal Investigator — Director of the International School of Aesthetic Medicine of the Fatebenefratelli Foundation
Locations (1):
- Fatebenefratelli Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araco A, Araco F. Preliminary Prospective and Randomized Study of Highly Purified Polynucleotide vs Placebo in Treatment of Moderate to Severe Acne Scars. Aesthet Surg J. 2021 Jun 14;41(7):NP866-NP874. doi: 10.1093/asj/sjab125. PMID 33755110